CLINICAL TRIAL: NCT01363765
Title: Pilot Roll Out of the Xpert MTB/Rif for the Diagnosis of Pulmonary Tuberculosis in Two Municipalities in Brazil: a Stepped Wedge Trial
Brief Title: Xpert MTB/Rif, a New Tool for the Diagnosis of Pulmonary Tuberculosis in Two Municipalities in Brazil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataulpho de Paiva Foundation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPPGH5254; GH5254 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2011-05-27; First posted 2011-06-02 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Tuberculosis
Keywords: diagnosis; polymerase chain reaction; sputum smear; stepped-wedge design; cost-effectiveness; Xpert MTB/Rif
MeSH Terms: conditions — Tuberculosis; Disease | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xpert MTB/Rif (Experimental): Sputum specimens arriving during intervention period will be submitted to this technology, a real-time automated polymerase chain reaction test
  Interventions: Other: Xpert MTB/Rif
- Sputum smear (Active Comparator): Sputum smears arriving in the laboratory during the observation period will be submitted to the classic routine smear staining
  Interventions: Other: Smear microscopy

INTERVENTIONS:
Other: Xpert MTB/Rif — Automatized RT-PCR for the detection of Mycobacterium tuberculosis, the agent of TB, in sputum samples
  Other Names: Intervention period
  Arms: Xpert MTB/Rif
Other: Smear microscopy — Sputum smears arriving in the laboratory during the observation period will be submitted to the classic routine smear staining. This would be the non-intervention (control) arm.
  Other Names: Observation
  Arms: Sputum smear

SUMMARY:
Diagnosis of tuberculosis (TB) is a challenge because sputum smear, the most rapid and inexpensive test, often fails to detect the disease, in around 20 to 30% of cases. Culture of sputum yields a correct diagnosis in up to 90% of cases, but results are only available in 4 to 8 weeks, depending on the method. A new test (Xpert MTB/Rif) based on a rapid technique, named polymerase chain reaction (PCR), detects TB in less than 2 hours over 95% of cases, in addition to identification of cases resistant to certain drugs used to treat TB. The test is expensive, but several studies have demonstrated its accuracy, and since most steps are automatized, savings can be expected from human resources work. The aims of our study are (1) to evaluate this tool as a substitute test for sputum smears in routine conditions; (2) evaluate if it is cost-effective, meaning that effectiveness of the test may outweigh the extra cost, and (3) evaluate the acceptability of the test among patients and health care workers.

DETAILED DESCRIPTION:
The main study consisted of a group-randomized pragmatic trial following a stepped-wedge design. The GeneXpert machines will be installed in laboratories of the basic health units in Rio de Janeiro and Manaus, two cities with a high burden of the disease in Brazil. Doctors will prescribe routine tests in the clinics. When sputum specimens arrive in the laboratory, instead of performing smears, the Xpert MTB/Rif will be performed during the intervention period. If positive, a sputum smear will also be performed. The intervention period will be preceded by an observation period during which routine will be kept unchanged, i.e., only smears will be performed. The observation period will serve as a comparator (control). The investigators will then see how many more cases were detected during the intervention period, and in particular, how many smear-negative cases were detected, compared to the observation period.

A total of 35,000 specimens are expected to be tested with the new technology in 14 laboratories. Laboratories, not individuals, will be randomized.

ELIGIBILITY:
Inclusion Criteria:

laboratories -and not subjects - will be randomized. All laboratories will start doing smears, when indicated by randomization, they will switch to Xpert MTB/Rif. There are no inclusion or exclusion criteria for the labs. Sputum specimens from non-diagnostic (follow up) patients, second samples for diagnostic tests, insufficient volume/visible blood specimens will be excluded from the Xpert testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34758 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Cobelens, MD, PhD, Study Chair — AIGHD Foundation and Department of Global Health, Academic Medical Center, University of Amsterdam
Locations (1):
- Laboratories of Rio de Janeiro Health Department, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Trajman A, Durovni B, Saraceni V, Menezes A, Cordeiro-Santos M, Cobelens F, Van den Hof S. Impact on Patients' Treatment Outcomes of XpertMTB/RIF Implementation for the Diagnosis of Tuberculosis: Follow-Up of a Stepped-Wedge Randomized Clinical Trial. PLoS One. 2015 Apr 27;10(4):e0123252. doi: 10.1371/journal.pone.0123252. eCollection 2015. PMID 25915745
- [Derived] Durovni B, Saraceni V, van den Hof S, Trajman A, Cordeiro-Santos M, Cavalcante S, Menezes A, Cobelens F. Impact of replacing smear microscopy with Xpert MTB/RIF for diagnosing tuberculosis in Brazil: a stepped-wedge cluster-randomized trial. PLoS Med. 2014 Dec 9;11(12):e1001766. doi: 10.1371/journal.pmed.1001766. eCollection 2014 Dec. PMID 25490549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Feb 4 to Oct 4 2012, all 11 primary care laboratories in Rio de Janeiro and 3 labs covering 70% of PTB diagnosis in Manaus participated. Over the same period, 4,660 patients were notified with PTB to SINAN (disease information database). Of these, 2,745 (59%) could be linked to test results in GAL (lab information system).
Pre-assignment Details: Samples (and not patients) were included if it was a first diagnostic sample in the intervention arm. Follow up (non diagnostic) samples were excluded for both arms, as were inadequate samples (insufficient material, blood stained-specimens) in the intervention group.
Groups:
- Xpert MTB/Rif: Sputum specimens arriving during intervention period were submitted to this technology, a real-time automated polymerase chain reaction test
- Sputum Smear: Sputum smears arriving in the laboratory during the observation period were submitted to the classic routine AFB smear staining, as per national guidelines. Two smears were requested.
Period: Overall Study
Arm/Group | Xpert MTB/Rif | Sputum Smear
Started | 18322 (This is number of participants enrolled, each with one sample submitted to Xpert in intervention arm) | 16436 (This is number of participants enrolled, each with one sample considered in baseline arm.)
Completed | 12522 (Excluded were duplicates, non-residents, missing age, unavailability of system (smears done instead)) | 11705 (Samples contributing to observation arm. Excluded were duplicates, non-residents, missing age.)
Not Completed | 5800 | 4731
Not completed — non-diagnostic | 2621 | 1124
Not completed — duplicate records | 736 | 3177
Not completed — non-resident | 156 | 76
Not completed — age not recorded (used for cross-linkage | 117 | 354
Not completed — smear during intervention | 2170 | 0

BASELINE CHARACTERISTICS:
Population: Those are notified patients with pulmonary TB by the clinics which drain to the 14 participant labs all participants who were notified whether or not they were linked to the lab database. Further analyses do not correspond to all notified patients, it included only those linked in both databases.
Groups:
- Xpert MTB/Rif: One sample of sputum specimens arriving during intervention period were submitted to this technology instead, a real-time automated polymerase chain reaction test
- Total: Total of all reporting groups
Arm/Group | Xpert MTB/Rif | Sputum Smear | Total
Number analyzed (Participants) | 2610 | 2050 | 4660
Age, Customized [Number; unit: participants]
  Between 15 and 39 years | 1395 | 1068 | 2463
  Between 40 and 59 years | 835 | 682 | 1517
  >=60 years | 324 | 244 | 568
  <=14 years | 56 | 56 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 928 | 736 | 1664
  Male | 1682 | 1314 | 2996
Region of Enrollment [Number; unit: participants]
  Brazil | 2610 | 2050 | 4660

OUTCOME MEASURES:

1. Primary Outcome: Notification Rate Ratio
Description: Proportion of additional bacteriologically confirmed notified TB cases during intervention period compared to the observation period Patients notified who had a positive test result. The notification rate (NR, i.e., number of notifications/100,000 population/year) ratio (NRR) is defined as the NR in the intervention period/NR in the observation period, and is presented in the statistical analysis section.
Time Frame: October 2012 (up to 2 years)
Population: Only patients found both in laboratory and in the notification databases were included since this is an outcome based on notification rates. Population growth during time was estimated. NR per 100,000 population
Measure: Number (95% Confidence Interval); unit: notifications/100,000 persons/year
Groups:
- Xpert MTB/Rif: One sample of sputum specimens arriving during intervention period was submitted to this technology
- Sputum Smear: Sputum smears arriving in the laboratory during the observation period were submitted to the classic routine smear staining
Arm/Group | Xpert MTB/Rif | Sputum Smear
Number analyzed (Participants) | 1385 | 831
notifications/100,000 persons/year | 48.7 [41.5 to 55.8] | 30.5 [24.9 to 36.1]
Statistical Analysis 1: Comparison: Xpert MTB/Rif vs Sputum Smear; cluster-averaged NNR=1.59 (CI95% 1.31-1.88) Absolute numbers informed in table do not allow calculation of notification rates; they are based on population size, not in total numbers and percentages; Test type: Superiority or Other; p < 0.01, Clustered Avareged — NR were calculated using an aggregated database consisting of 896 strata for laboratory (n=14), study month (n=8), sex (n=2) and age group (n=4: <15, 15-39, 40-59, and >=60 years). Poisson regression modeling was used to analyze changes in TB TB NR; Adjustment for municipality, age, sex, and baseline proportion of samples with a positive smear was by a population-averaged quasi-likelihood approach; notification rate ratio = 1.59, 95% CI 2-sided [1.32 to 1.87] — The numbers reported in the "CONSORT" flowchart refer to the diagnostic samples. NR were obtained crosslinking lab and notification databases, denominator was population/year
Statistical Analysis 2: Comparison: Xpert MTB/Rif vs Sputum Smear; Secondary analysis: Mixed multi-level model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mixed multi-level model, time-adjusted; notification rate ratio = 1.70, 95% CI 2-sided [1.51 to 1.92]

2. Primary Outcome: Costs Per Detected Case
Description: Costs per detected case were analyzed using a decision tree model from the national health system perspective. Incremental cost-effectiveness ratio (ICER) was calculated as (costs with Xpert - costs with smears)/(cases detected with Xpert - cases detected with smears). Negative ICERs mean cost saving.
Time Frame: October 2012 (up to 2 years)
Measure: Number; unit: American dollars
Arm/Group | Xpert MTB/Rif | Sputum Smear
Number analyzed (Participants) | 12522 | 11705
American dollars | 714.95 | 799.02
Statistical Analysis 1: Comparison: Xpert MTB/Rif vs Sputum Smear; Test type: Superiority or Other; Incremental cost-effectiveness ratio (ICER) per case detected; incremental cost-effectiveness ratio = -84.07

3. Secondary Outcome: NRR of Non-laboratory Tested TB (Cluster-averaged).
Description: The notification rate (NR, i.e., number of notifications/100,000 population/year) ratio (NRR) is defined as the NR in the intervention period/NR in the observation period, and is presented in the statistical analysis section.
  Numbers are participants in the notification database who were not in the lab (all tests done) database; denominators are population taking into account growth of the population during the study period, adjusted for variations in monthly number of opening days (by weighing the number of person-months for the proportion of suspects with samples examined each month out of the total number examined by the laboratory during the whole study period), stratified by sex and age group.
  Routine practices were not changed; patients with a high suspicion of TB were, as prior to the study, notified regardless of a confirmatory test.
Time Frame: October 2012 (up to 2 years)
Population: The result is the notification rate ratio
Measure: Number (95% Confidence Interval); unit: notifications/100,000 persons/year
Arm/Group | Xpert MTB/Rif | Sputum Smear
Number analyzed (Participants) | 1009 | 906
notifications/100,000 persons/year | 35.8 [27.6 to 43.9] | 36.9 [26.8 to 47.1]
Statistical Analysis 1: Comparison: Xpert MTB/Rif vs Sputum Smear; Test type: Superiority or Other; p = 0.923, Agregated cluster-averaged — cluster-averaged adjusted NRR (notification rate ratio, not calculable from number shown, which are a proportion of tests. NRR calculated over a population/year denominator; NRR = 0.98, 95% CI 2-sided [0.64 to 1.32]

4. Secondary Outcome: NRR of Negative-laboratory TB (Cluster-averaged).
Description: The notification rate (NR, i.e., number of notifications/100,000 population/year) ratio (NRR) is defined as the NR in the intervention period/NR in the observation period, and is presented in the statistical analysis section.
  Numbers are driven from linkage between lab (all tests done) and notification databases; denominators are population taking into account growth of the population during the study period, adjusted for variations in monthly number of opening days (by weighing the number of person-months for the proportion of suspects with samples examined each month out of the total number examined by the laboratory during the whole study period), stratified by sex and age group.
  Routine practices were not changed; patients with a high suspicion of TB were, as prior to the study, notified regardless of a confirmatory test.
Time Frame: October 2012 (up to 2 years)
Measure: Number (95% Confidence Interval); unit: notifications/100,000 persons/year
Arm/Group | Xpert MTB/Rif | Sputum Smear
Number analyzed (Participants) | 216 | 313
notifications/100,000 persons/year | 7.3 [2.1 to 12.5] | 12.1 [6.1 to 18.0]
Statistical Analysis 1: Comparison: Xpert MTB/Rif vs Sputum Smear; Test type: Superiority or Other; p = 0.004, Agregated cluster-averaged — cluster-averaged adjusted NRR; NRR = 0.52, 95% CI 2-sided [0.21 to 0.84]

ADVERSE EVENTS:
Description: Serious and Other (non-serious) Adverse Events were not collected/assessed
Arm/Group | Xpert MTB/Rif | Sputum Smear
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The design has potential for bias, due to delayed treatment effects or to conditions that change over time. Both are unlikely: outcome (notification) was shortly after test and adjustment for time in multilevel mixed model confirmed primary analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No